CLINICAL TRIAL: NCT00416637
Title: Biomarker and Clinical Evaluation of Bevacizumab (Avastin) to Determine the Role of Nitric Oxide in Anti-VEGF Therapy
Brief Title: Bevacizumab in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Herbert Hurwitz, MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Herbert Hurwitz, MD, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00008011; DUMC-4907-05-6R2; GENENTECH-DUMC-4907-05-6R2; CDR0000449969 (Other: NCI)
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Bevacizumab

ARMS (1):
- Bevacizumab (Avastin) (Experimental): Bevacizumab given and then BP checked and skin biopsies obtained.
  Interventions: Biological: Bevacizumab (Avastin)

INTERVENTIONS:
Biological: Bevacizumab (Avastin)

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some find tumor cells and kill them or carry tumor-killing substances to them. Others interfere with the ability of tumor cells to grow and spread. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor .

PURPOSE: This phase I trial is studying how well bevacizumab works in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether anti-vascular epidermal growth factor (VEGF) treatment comprising bevacizumab causes changes in endothelial cell function, as measured by brachial reactivity, and changes in nitric oxide (NOx), as measured by plasma/urinary/exhaled NOx levels, in patients with advanced solid tumors.
* Determine whether anti-VEGF-related changes in blood pressure correlate with changes in brachial reactivity and NOx levels.

Secondary

* Evaluate anti-angiogenic effects of bevacizumab in neovascular tissue in the wound angiogenesis model.
* Correlate inhibition of wound angiogenesis with changes in VEGF-receptor 2 phosphorylation status and changes in NOx synthase expression.
* Describe the mean and associated variability of other plasma and urine markers known to be associated with vascular reactivity, endothelial function, and/or tumor angiogenesis.
* Describe, preliminarily, whether these changes correlate with changes in blood pressure, brachial reactivity, NOx levels, or wound angiogenesis.

OUTLINE: Patients receive bevacizumab IV over 30-90 minutes on days 1, 15, and 29. After the third dose of bevacizumab, patients may receive additional bevacizumab in combination with chemotherapy in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumor

  * Metastatic or unresectable disease
* Standard curative or palliative measures do not exist or are no longer effective OR treatment with standard chemotherapy plus bevacizumab is appropriate* NOTE: *It must be judged clinically appropriate by the treating physician to delay combination treatment for the 6 weeks needed for study participation
* Patients with squamous cell non-small cell lung cancer are ineligible

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute neutrophil count ≥ 2,000/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9.0 g/dL
* AST/ALT ≤ 2.5 times upper limit of normal (ULN) (5 times ULN if known liver metastases are present)
* Creatinine clearance ≥ 50 mL/min
* No proteinuria at baseline

  * Patients with ≥ 1+ proteinuria during screening should undergo a timed 12- or 24-hour urine collection, which must be an adequate collection and must demonstrate < 500 mg protein/24 hr to be eligible for the study
* Not pregnant or nursing

  * No nursing for ≥ 4 months after completion of study treatment
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 4 months after completion of study treatment
* No arterial thromboembolic events within the past 6 months, including any of the following:

  * Transient ischemic attack
  * Cerebrovascular accident
  * Unstable angina
  * Myocardial infarction
  * Clinically significant peripheral vascular disease
* No venous thromboembolic event within the past 3 months
* No clinically significant cardiovascular disease
* No uncontrolled hypertension
* No New York Heart Association class II or greater congestive heart failure
* No serious cardiac arrhythmia requiring medication

  * Atrial or supraventricular tachycardias that are well controlled with beta blockers or calcium channel blockers are allowed
  * Chronic pacemakers allowed
* No presence of bleeding diathesis or coagulopathy
* No significant traumatic injury within the past 4 weeks
* No history of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the patient at high risk from treatment complications

PRIOR CONCURRENT THERAPY:

* No administration of nitrates within the past week
* At least 2 weeks since prior and no concurrent antihypertensive agent(s)

  * Must have stable blood pressure (BP) (BP < 160/100 mm Hg) within the past 2 weeks
  * Must be asymptomatic within the past 2 weeks
* No open biopsy within the past 14 days
* No fine needle aspirations other than in the breast within the past 7 days
* No placement of a vascular access device within the past 7 days
* No major surgical procedure within the past 4 weeks
* No chemotherapy within the past 4 weeks (6 weeks for nitrosoureas or mitomycin C) and recovered
* No radiotherapy within the past 4 weeks
* No previous treatment with bevacizumab
* No need for major surgical procedure during the course of the study
* No other cancer immunotherapy or biologic therapy while on the study
* No concurrent or recent (within past 10 days) use of full-dose oral or parenteral anticoagulants (heparin > 10,000/day or an INR > 1.5) or thrombolytic agents

  * 1 mg of warfarin is permitted as required to maintain patency of preexisting, permanent indwelling IV catheters
* No chronic, daily treatment with aspirin (> 325 mg/day) or nonsteroidal anti-inflammatory medications (of the kind known to inhibit platelet function at doses used to treat chronic inflammatory diseases)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2004-01; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert I. Hurwitz, MD, Principal Investigator — Duke Cancer Institute